CLINICAL TRIAL: NCT00208351
Title: Clinical and Radiographic Evaluation to Compare a Polished and Non-polished Collared Stem and a Polished and Non Polished Collarless Stem in Primary Total Hip Replacement
Brief Title: A Randomised Single Centre Study to Compare the Long-term Performance of 4 Designs of the DePuy Ultima LX Stem in Primary Total Hip Replacement
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The final assessments were conducted late and in a reduced format due to resource limitations at the site.
Sponsor: DePuy International (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CT01/95
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2016-05-11 (Estimated); Status verified 2016-03

CONDITIONS: Osteoarthritis; Post-traumatic Arthritis; Collagen Disorder; Avascular Necrosis; Traumatic Femoral Fractures; Nonunion of Femoral Fractures; Congenital Hip Dysplasia; Slipped Capital Femoral Epiphysis
Keywords: Hip; Cemented
MeSH Terms: conditions — Osteoarthritis; Collagen Diseases; Osteonecrosis; Hip Dislocation, Congenital; Slipped Capital Femoral Epiphyses

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1) Ultima LX Collared Stem - Non-Polished/Blasted Finished (Active Comparator): A collared non-polished blasted finished cementless femoral component for use in total hip replacement.
  Interventions: Device: Ultima LX Collared Stem - Non-Polished/Blasted Finished
- 2) Ultima LX Collared Stem - Polished Finished (Active Comparator): A collared polished finished cementless femoral component for use in total hip replacement.
  Interventions: Device: Ultima LX Collared Stem - Polished Finished
- 3) Ultima LX Collarless Stem - Non-Polished/Blasted Finished (Active Comparator): A collarless non-polished/blasted finished cementless femoral component for use in total hip replacement.
  Interventions: Device: Ultima LX Collarless Stem - Non-Polished/Blasted Finished
- 4) Ultima LX Collarless Stem - Polished Finished (Active Comparator): A collarless polished finished cementless femoral component for use in total hip replacement.
  Interventions: Device: Ultima LX Collarless Stem - Polished finished

INTERVENTIONS:
Device: Ultima LX Collared Stem - Non-Polished/Blasted Finished — A collared non-polished/blasted finished cementless femoral component for use in total hip replacement.
  Arms: 1) Ultima LX Collared Stem - Non-Polished/Blasted Finished
Device: Ultima LX Collared Stem - Polished Finished — A collared polished finished cementless femoral component for use in total hip replacement.
  Arms: 2) Ultima LX Collared Stem - Polished Finished
Device: Ultima LX Collarless Stem - Non-Polished/Blasted Finished — A collarless non-polished/blasted finished cementless femoral component for use in total hip replacement.
  Arms: 3) Ultima LX Collarless Stem - Non-Polished/Blasted Finished
Device: Ultima LX Collarless Stem - Polished finished — A collarless polished finished cementless femoral component for use in total hip replacement.
  Arms: 4) Ultima LX Collarless Stem - Polished Finished

SUMMARY:
The purpose of this study is to compare the performance of 4 designs of the DePuy Ultima LX hip stem in the treatment of patients with hip joint disease requiring a total hip replacement. Patients who enter the study will be randomly allocated to one of the 4 designs of the DePuy Ultima LX hip stem and will be evaluated at regular intervals following hip surgery using patient, clinical and x-ray assessments.

ELIGIBILITY:
Inclusion Criteria:

Current indications for primary total hip arthroplasty utilising a cemented femoral component. These include pain, deformity and loss of function which are not responsive to medical treatment

Exclusion Criteria:

i) Revision Total Hip Arthroplasty ii) Rheumatoid arthritis iii) Age greater than 80 years at time of surgery iv) Age less than 60 years at time of surgery v) Previous hip joint sepsis vi) Obesity vii) Patient likely to remain housebound once rehabilitation is complete

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 1997-05; Primary Completion 2004-11 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Stem movement measured radiographically at 2 years | 2yrs post-surgery
  Stem movement was measured radiographically by comparing baseline stem position with the stem position 2 years after surgery. If migration was observed to be 5 or more mm, it was considered clinically significant migration.

SECONDARY OUTCOMES:
Comparisons of Visual Analog Pain (VAS), 36-Item Short Form Health Survey (SF-36), Satisfaction, Limb Length and stem movement measured radiographically at 5 years. | 5yrs post-surgery
  The following outcome measures were used; VAS Pain score, SF36 Patient reported outcome, Satisfaction, Limb Length physical examination, and stem movement measured radiographically.

CONTACTS AND LOCATIONS:
Locations (1):
- Epsom General Hospital, Surrey, United Kingdom

REFERENCES:
- [Result] Hutt J, Hazlerigg A, Aneel A, Epie G, Dabis H, Twyman R, Cobb A. The effect of a collar and surface finish on cemented femoral stems: a prospective randomised trial of four stem designs. Int Orthop. 2014 Jun;38(6):1131-7. doi: 10.1007/s00264-013-2256-z. Epub 2014 Jan 29. PMID 24474088